CLINICAL TRIAL: NCT04660838
Title: Intervention to REduce anticholinerGic burdEN in oldER pATiEnts (REGENERATE) Aged 65 Years and Older: A Non-randomised Feasibility Study
Brief Title: Intervention to REduce anticholinerGic burdEN in oldER pATiEnts (REGENERATE) Aged 65 Years and Older
Acronym: REGENERATE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2-094-20
Record Dates: First submitted 2020-12-01; First posted 2020-12-09 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Anticholinergic Adverse Reaction
Keywords: Anticholinergic burden

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: ACB intervention — Stopping and/or switching ACB medication to an alternative
  Other Names: Stopping and/or switching ACB medication

SUMMARY:
Medications with anticholinergic properties are frequently prescribed for several conditions in older age; for example cardiovascular drugs (e.g. digoxin, furosemide), urologicals (e.g. darifenacin, oxybutynin) and anti-parkinsonism drugs (e.g. benztropine, trihexyphenadyl). It has been shown that increasing anticholinergic burden (ACB) can cause poor health-related outcomes, but there are still uncertainties around whether it is possible or acceptable to stop medication with high ACB and/or switching to another medication with no or low anticholinergic burden, the effect on health-related outcomes of such an approach, the most appropriate person to deliver this intervention or the health care setting in which it should take place.

The term 'deprescribing' is the process of intentionally stopping a medication or reducing its dose to improve the person's health or reduce the risk of adverse side effects. There is, however, limited research regarding deprescribing. Previously, researchers have suggested deprescribing is a systematic process of identifying and discontinuing drugs in instances in which existing or potential harms outweigh existing or potential benefits within the context of an individual patient's care goals, current level of functioning, life expectancy, values, and preferences. However, there are not many studies about implementation of appropriate interventions to reduce ACB in older patients (aged 65 year and over).

The aim of this non-randomised study is to explore the feasibility of delivering an intervention to reduce the ACB in older patients by deprescribing or switching to inform a future definitive clinical trial. This is a single-arm, open feasibility study conducted in primary and secondary care involving older patients. Mixed method (routine data, questionnaires and interviews) will be used in this study.

ELIGIBILITY:
Inclusion Criteria for stopping and/or switching medications

Patients who are:

* aged 65 and over
* able to provide informed consent.
* on one or more long-term drugs (have been prescribed a minimum 6 weeks) with ACB potential (Anticholinergic Cognitive Burden scale ≥3) (defined according to Boustani et al (Boustani, Campbell et al. 2008)

Exclusion Criteria for stopping and/or switching medications

Patients who:

* are without capacity to provide informed consent.
* have severe mental illness [such as diagnosis of severe anxiety, severe depression, severe dementia etc.].
* are terminally ill (life expectancy less than 6 months).
* in opinion of responsible clinician are not suitable.
* are taking part in another study.

Health care professional inclusion criteria for interviews

- Professionals: doctors (consultants, GPs), pharmacist in primary and secondary care involved in the care of patients aged 65 and over on polypharmacy regimes/likely to have anticholinergic burden and have taken part in the study by delivering the intervention

Patients inclusion criteria for interviews

- Patients: patients aged 65 years and over who met eligible criteria and have taken part in the REGENERATE study will be selected.

Exclusion criteria for interviews

- Participants who cannot understand English fluently

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-07-17 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Recruitment of patients from GP practices and hospitals | 3 months
  The number of patients who are invited to study and the number of patients agree to take part and refuse with reasons.
The completion rate of baseline and follow up data | 3 months
  The patients background information, medical history, medications will be recorded at baseline and at 3 months.
The number of medication changes recommended and the number implemented | 3 months
  Time taken to do consultations and acceptance as well as rejection with reasons of doctor from pharmacist recommendations.
The sustainability of intervention (i.e. those remained on same drugs at 6 week and 3 months post intervention) | 3 months
  Information on patients who remained on reduced regimen and those who went back on the drug or need extra-drug and reasons.
The acceptability of intervention to patients and health care professional stakeholders | 3 months
  Semi-structured interviews with patients and health care professionals

CONTACTS AND LOCATIONS:
Locations (1):
- Peterculter Medical Practice, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Best O, Gnjidic D, Hilmer SN, Naganathan V, McLachlan AJ. Investigating polypharmacy and drug burden index in hospitalised older people. Intern Med J. 2013 Aug;43(8):912-8. doi: 10.1111/imj.12203. PMID 23734965
- [Background] BOUSTANI, M., CAMPBELL, N., MUNGER, S., MAIDMENT, I. and FOX, C., 2008. Impact of anticholinergics on the ageing brain: a review and practical application. Aging Health, 4(3), pp. 311-320.
- [Background] Cancelli I, Beltrame M, Gigli GL, Valente M. Drugs with anticholinergic properties: cognitive and neuropsychiatric side-effects in elderly patients. Neurol Sci. 2009 Apr;30(2):87-92. doi: 10.1007/s10072-009-0033-y. Epub 2009 Feb 20. PMID 19229475
- [Background] Feinberg M. The problems of anticholinergic adverse effects in older patients. Drugs Aging. 1993 Jul-Aug;3(4):335-48. doi: 10.2165/00002512-199303040-00004. PMID 8369593
- [Background] Fox C, Smith T, Maidment I, Chan WY, Bua N, Myint PK, Boustani M, Kwok CS, Glover M, Koopmans I, Campbell N. Effect of medications with anti-cholinergic properties on cognitive function, delirium, physical function and mortality: a systematic review. Age Ageing. 2014 Sep;43(5):604-15. doi: 10.1093/ageing/afu096. Epub 2014 Jul 19. PMID 25038833
- [Background] Gorup E, Rifel J, Petek Ster M. Anticholinergic Burden and Most Common Anticholinergic-acting Medicines in Older General Practice Patients. Zdr Varst. 2018 Jun 21;57(3):140-147. doi: 10.2478/sjph-2018-0018. eCollection 2018 Jun. PMID 29983780
- [Background] Green AR, Reifler LM, Bayliss EA, Weffald LA, Boyd CM. Drugs Contributing to Anticholinergic Burden and Risk of Fall or Fall-Related Injury among Older Adults with Mild Cognitive Impairment, Dementia and Multiple Chronic Conditions: A Retrospective Cohort Study. Drugs Aging. 2019 Mar;36(3):289-297. doi: 10.1007/s40266-018-00630-z. PMID 30652263
- [Background] Kersten H, Molden E, Tolo IK, Skovlund E, Engedal K, Wyller TB. Cognitive effects of reducing anticholinergic drug burden in a frail elderly population: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2013 Mar;68(3):271-8. doi: 10.1093/gerona/gls176. Epub 2012 Sep 14. PMID 22982689
- [Background] Lopez-Alvarez J, Sevilla-Llewellyn-Jones J, Aguera-Ortiz L. Anticholinergic Drugs in Geriatric Psychopharmacology. Front Neurosci. 2019 Dec 6;13:1309. doi: 10.3389/fnins.2019.01309. eCollection 2019. PMID 31866817
- [Background] Nakham A, Myint PK, Bond CM, Newlands R, Loke YK, Cruickshank M. Interventions to Reduce Anticholinergic Burden in Adults Aged 65 and Older: A Systematic Review. J Am Med Dir Assoc. 2020 Feb;21(2):172-180.e5. doi: 10.1016/j.jamda.2019.06.001. Epub 2019 Jul 24. PMID 31351858
- [Background] OLASEHINDE-WILLIAMS, O., July, 2020-last update, Deprescribing guide. Available: https://southendccg.nhs.uk/your-health-services/healthcare-professionals/medicines-management/medicines-management-resources/2308-deprescribing-guide/file [April/03, 2020].
- [Background] Reeve E, Shakib S, Hendrix I, Roberts MS, Wiese MD. The benefits and harms of deprescribing. Med J Aust. 2014 Oct 6;201(7):386-9. doi: 10.5694/mja13.00200. PMID 25296058